CLINICAL TRIAL: NCT05393869
Title: The Effect of Nicotine and Tobacco Message Framing on Use Among Diverse Groups of Young Adults
Brief Title: Evaluating Anti-Tobacco Message Effectiveness Among Lesbian, Gay, Bisexual, and Transgender Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Joanne Patterson, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: OSU-20427; NCI-2022-02543 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); K99CA260718 (NIH)
Record Dates: First submitted 2022-05-18; First posted 2022-05-26 (Actual); Results first posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Tobacco-Related Carcinoma
MeSH Terms: interventions — Health Communication

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- AR-Quit (Experimental): Participants view messages with absolute risk and quit statements
  Interventions: Other: Health communications
- AR-Switch (Experimental): Participants view messages with absolute risk and switch statements
  Interventions: Other: Health communications
- AR-Combination (Experimental): Participants view messages with absolute risk and combination quit+switch statements
  Interventions: Other: Health communications
- RR-Quit (Experimental): Participants view messages with comparative risk and quit statements
  Interventions: Other: Health communications
- RR-Switch (Experimental): Participants view messages with comparative risk and switch statements
  Interventions: Other: Health communications
- RR-Combination (Experimental): Participants view messages with comparative risk and combination quit+switch statements
  Interventions: Other: Health communications
- Control (Other): Participants view FDA regulatory messages
  Interventions: Other: Health communications

INTERVENTIONS:
Other: Health communications — Participants are assigned to view health communications with risk and efficacy statements.

SUMMARY:
This trial refines and evaluates anti-tobacco messages among lesbian, gay, bisexual, and transgender (LGBT) young adults at risk for the use of more than one tobacco product (polytobacco use). Polytobacco use is associated with nicotine dependence and tobacco use into adulthood, and is disproportionately high among LGBT young adults. This trial seeks to determine effective communication of polytobacco use risk to at-risk LGBT young adults.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Identify absolute and relative risk anti-tobacco messages that effectively communicate polytobacco risks to lesbian, gay, bisexual, transgender (LGBT) young adults.

Participants view anti-tobacco messages and rate them for perceived effectiveness and reactance.

ELIGIBILITY:
Inclusion Criteria:

* Young adults (age 18-35 years)
* Live in the United States

At least 50% of the sample also:

* Are susceptible to multiple nicotine and tobacco product use (i.e., have used combustible tobacco or e-cigarettes at least once)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2849 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne G Patterson, PhD MPH MSW, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AR-Quit | AR-Switch | AR-Combination | RR-Quit | RR-Switch | RR-Combination | Control
Started | 407 | 407 | 407 | 407 | 407 | 407 | 407
Completed | 400 | 405 | 398 | 404 | 402 | 403 | 404
Not Completed | 7 | 2 | 9 | 3 | 5 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AR-Quit | AR-Switch | AR-Combination | RR-Quit | RR-Switch | RR-Combination | Control | Total
Number analyzed (Participants) | 407 | 407 | 407 | 407 | 407 | 407 | 407 | 2849
Age, Customized [Count of Participants; unit: Participants]
  18-24 years old | 131 | 123 | 138 | 126 | 133 | 139 | 138 | 928
  25-35 years old | 270 | 283 | 261 | 278 | 270 | 265 | 267 | 1894
  Unknown or not reported | 6 | 1 | 8 | 3 | 4 | 3 | 2 | 27
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Cisgender female | 195 | 192 | 195 | 187 | 224 | 187 | 185 | 1365
  Cisgender Male | 169 | 183 | 163 | 179 | 152 | 171 | 180 | 1197
  Transgender or gender diverse | 36 | 30 | 41 | 38 | 27 | 46 | 40 | 258
  Unknown or not reported | 7 | 2 | 8 | 3 | 4 | 3 | 2 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 58 | 59 | 49 | 57 | 45 | 62 | 48 | 378
  Not Hispanic or Latino | 343 | 347 | 350 | 347 | 358 | 342 | 357 | 2444
  Unknown or Not Reported | 6 | 1 | 8 | 3 | 4 | 3 | 2 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 4 | 3 | 4 | 4 | 2 | 22
  Asian | 30 | 39 | 28 | 43 | 31 | 36 | 31 | 238
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 5
  Black or African American | 47 | 41 | 45 | 39 | 42 | 55 | 53 | 322
  White | 253 | 256 | 258 | 246 | 266 | 244 | 264 | 1787
  More than one race | 24 | 24 | 29 | 32 | 32 | 27 | 16 | 184
  Unknown or Not Reported | 50 | 45 | 42 | 43 | 31 | 41 | 39 | 291
Region of Enrollment [Number; unit: participants]
  United States | 407 | 407 | 407 | 407 | 407 | 407 | 407 | 2849
Sexual Orientation [Count of Participants; unit: Participants]
  Heterosexual | 206 | 225 | 200 | 215 | 215 | 220 | 212 | 1493
  Lesbian or gay | 46 | 43 | 38 | 45 | 37 | 46 | 44 | 299
  Bisexual | 129 | 121 | 131 | 126 | 141 | 124 | 133 | 905
  Ace/Asexual | 19 | 17 | 29 | 16 | 10 | 13 | 14 | 118
  Unknown or not reported | 7 | 1 | 9 | 5 | 4 | 4 | 4 | 34
Smoking status [Count of Participants; unit: Participants] — Participants self-identified as currently using combustible cigarettes (use within the past 30-days), formerly using cigarettes (used at least once in lifetime, but not within past 30-days), and never using cigarettes.
  Participants
    Currently use cigarettes | 108 | 114 | 106 | 106 | 93 | 106 | 117 | 750
    Formerly used cigarettes | 168 | 148 | 176 | 170 | 192 | 171 | 159 | 1184
    Never used cigarettes | 131 | 145 | 125 | 131 | 122 | 130 | 131 | 915
    Unknown or not reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaping status [Count of Participants; unit: Participants] — Participants self-identified as currently using nicotine vapes (use within the past 30-days), formerly using nicotine vapes (used at least once in lifetime, but not within past 30-days), and never using nicotine vapes.
  Participants
    Currently vape nicotine | 141 | 144 | 146 | 137 | 160 | 147 | 140 | 1015
    Formerly vaped nicotine | 139 | 133 | 132 | 141 | 118 | 117 | 135 | 915
    Never vaped nicotine | 127 | 130 | 129 | 129 | 129 | 143 | 132 | 919
    Unknown or not reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dual smoking/vaping status [Count of Participants; unit: Participants] — Participants self-identified as currently using both combustible cigarettes and nicotine vapes (use within the past 30-days), formerly using both cigarettes and nicotine vapes (used at least once in lifetime, but not within past 30-days), currently using cigarettes OR nicotine vapes (not both), or never using either cigarettes or nicotine vapes.
  Participants
    Currently vape nicotine AND smoke cigarettes | 63 | 73 | 65 | 57 | 61 | 64 | 69 | 452
    Formerly vaped nicotine AND smoked cigarettes | 177 | 162 | 176 | 177 | 184 | 169 | 168 | 1213
    Only ever vaped nicotine OR smoked cigarettes | 76 | 69 | 78 | 86 | 73 | 75 | 77 | 534
    Never vaped nicotine OR smoked cigarettes | 91 | 103 | 88 | 87 | 89 | 99 | 93 | 650
    Unknown or not reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Message Perceived Effectiveness - Persuasive Potential.
Description: 6 items measured on 5-point scale, 1 = Not at all and 5 = Very much
  * These messages were worth remembering.
  * These messages grabbed my attention.
  * These messages are powerful.
  * These messages are convincing.
  * These messages are meaningful.
  * These messages are informative.
  Responses were summed and averaged to create a scale for intention to quit (range from 1 - 5).
  Higher scores indicate a higher persuasive potential of the message.
Time Frame: Immediately post-exposure to intervention, up to 1 hour
Population: Analytic population only included participants who had no missing data for any scale items.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | AR-Quit | AR-Switch | AR-Combination | RR-Quit | RR-Switch | RR-Combination | Control
Number analyzed (Participants) | 399 | 402 | 396 | 403 | 401 | 402 | 402
units on a scale | 3.57 [3.47 to 3.67] | 3.24 [3.13 to 3.35] | 3.26 [3.15 to 3.36] | 3.44 [3.33 to 3.54] | 2.93 [2.42 to 3.44] | 2.98 [2.48 to 3.49] | 3.10 [2.96 to 3.24]

2. Primary Outcome: Perceived Effectiveness - Perceived Behavioral Impact
Description: Six items were analyzed separately, each scored on 5-point Likert scale (1=Strongly Disagree, 5=Strongly Agree)
  These messages will motivate CIGARETTE SMOKERS to switch to vaping.
  These messages will motivate people to quit ALL smoking and vaping.
  These messages will motivate NON-USERS to start vaping.
  These messages will motivate NON-USERS to start smoking cigarettes.
  These messages will motivate CIGARETTE SMOKERS to quit.
  These messages will motivate VAPERS to quit.
Time Frame: Immediately post-exposure to intervention, up to 1 hour
Population: Analytic population did not include participants with missing data for outcomes.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | AR-Quit | AR-Switch | AR-Combination | RR-Quit | RR-Switch | RR-Combination | Control
Number analyzed (Participants) | 403 | 407 | 399 | 405 | 403 | 405 | 405
units on a scale
  These messages will motivate people to quit ALL smoking and vaping. | 2.96 [2.84 to 3.08] | 2.38 [2.25 to 2.50] | 2.44 [2.32 to 2.56] | 2.71 [2.59 to 2.84] | 2.07 [1.96 to 2.19] | 2.22 [2.11 to 2.34] | 2.76 [2.63 to 2.88]
  These messages will motivate CIGARETTE SMOKERS to quit. | 3.11 [2.97 to 3.23] | 3.10 [2.98 to 3.22] | 3.16 [3.04 to 3.27] | 3.28 [3.17 to 3.40] | 3.00 [2.88 to 3.11] | 3.17 [3.04 to 3.29] | 2.82 [2.70 to 2.95]
  These messages will motivate CIGARETTE SMOKERS to switch to vaping | 2.10 [2.00 to 2.21] | 3.52 [3.40 to 3.63] | 3.41 [3.29 to 3.53] | 3.34 [3.22 to 3.45] | 3.67 [3.57 to 3.78] | 3.67 [3.56 to 3.78] | 1.81 [1.72 to 1.91]
  These messages will motivate VAPERS to quit. | 2.96 [2.84 to 3.08] | 2.21 [2.09 to 2.33] | 2.26 [2.14 to 2.37] | 2.53 [2.41 to 2.64] | 1.84 [1.73 to 1.94] | 1.94 [1.83 to 2.04] | 2.83 [2.71 to 2.95]
  These messages will motivate NON-USERS to start vaping. | 1.26 [1.20 to 1.33] | 1.91 [1.80 to 2.02] | 1.87 [1.75 to 1.98] | 1.62 [1.53 to 1.72] | 2.17 [2.05 to 2.29] | 2.14 [2.02 to 2.26] | 1.26 [1.20 to 1.33]
  These messages will motivate NON-USERS to start smoking cigarettes. | 1.24 [1.17 to 1.30] | 1.29 [1.22 to 1.36] | 1.35 [1.27 to 1.42] | 1.21 [1.15 to 1.27] | 1.30 [1.23 to 1.37] | 1.32 [1.25 to 1.40] | 1.24 [1.18 to 1.30]

3. Primary Outcome: Risk Perceptions: Absolute/Relative Risks of Cigarette vs. E-cigarette Use
Description: On a scale from 0-10, where 0 = not at all harmful and 10 = extremely harmful now harmful are ... to your health?
  * combustible cigarettes
  * nicotine vapes
  On a scale from 0-10, where 0 = much less harmful and 10 = much more harmful...
  • compared to combustible cigarettes, how harmful are nicotine vapes to your health?
Time Frame: Immediately post-exposure to intervention, up to 1 hour
Population: Analytic population included participants with no missing data on outcomes.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | AR-Quit | AR-Switch | AR-Combination | RR-Quit | RR-Switch | RR-Combination | Control
Number analyzed (Participants) | 399 | 402 | 396 | 403 | 402 | 402 | 403
units on a scale
  Absolute harm of cigarettes to health | 9.08 [8.95 to 9.21] | 9.07 [8.93 to 9.21] | 8.97 [8.82 to 9.12] | 9.11 [8.98 to 9.24] | 9.06 [8.93 to 9.20] | 9.04 [8.89 to 9.19] | 8.94 [8.79 to 9.09]
  Absolute harm of nicotine vapes to health | 7.57 [7.35 to 7.79] | 7.05 [6.83 to 7.27] | 7.19 [6.96 to 7.42] | 7.19 [6.97 to 7.42] | 6.88 [6.64 to 7.11] | 6.94 [6.71 to 7.17] | 7.57 [7.34 to 7.80]
  Relative harm of nicotine vapes (vs combustible cigarettes) to health | 4.99 [4.71 to 5.26] | 4.65 [4.38 to 4.92] | 4.81 [4.51 to 5.11] | 4.46 [4.16 to 4.75] | 4.34 [4.05 to 4.64] | 4.49 [4.20 to 4.78] | 5.04 [4.77 to 5.30]

4. Primary Outcome: Behavioral Intentions to Use Tobacco
Description: 8-items made up two 4-pt scales (1 = definitely will not and 4 = definitely will).
  Items for each scale were summed and averaged. Higher scores indicate higher likelihood of avoiding cigarettes/nicotine vapes.
  How likely it is that in the next 3 months, you will refrain from...
  * smoking cigarettes completely and permanently?
  * smoking cigarettes when you get lonely?
  * smoking cigarettes when you are with your friends who use them?
  * smoking cigarettes when someone hands you a cigarette?
  How likely it is that in the next 3 months, you will refrain from...
  * vaping nicotine completely and permanently?
  * vaping nicotine when you get lonely?
  * vaping nicotine when you are with your friends who use them?
  * vaping nicotine when someone hands you a vape?
Time Frame: Immediately post-exposure to intervention, up to 1 hour
Population: Analytic population included participants who did not have missing data on outcomes.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | AR-Quit | AR-Switch | AR-Combination | RR-Quit | RR-Switch | RR-Combination | Control
Number analyzed (Participants) | 403 | 407 | 399 | 405 | 403 | 405 | 405
units on a scale
  Behavioral intentions to use nicotine vapes | 3.27 [3.17 to 3.36] | 3.16 [3.06 to 3.26] | 3.16 [3.06 to 3.27] | 3.22 [3.12 to 3.31] | 3.11 [3.01 to 3.22] | 3.17 [3.07 to 3.27] | 3.15 [3.04 to 3.25]
  Behavioral intentions to smoke cigarettes | 3.48 [3.40 to 3.56] | 3.40 [3.31 to 3.49] | 3.40 [3.30 to 3.49] | 3.46 [3.37 to 3.54] | 3.46 [3.38 to 3.55] | 3.44 [3.35 to 3.52] | 3.37 [3.28 to 3.46]

ADVERSE EVENTS:
Time Frame: 1 hour post-baseline
Arm/Group | AR-Quit | AR-Switch | AR-Combination | RR-Quit | RR-Switch | RR-Combination | Control
All-Cause Mortality (participants affected / at risk) | 0/407 | 0/407 | 0/407 | 0/407 | 0/407 | 0/407 | 0/407
Serious Adverse Events (participants affected / at risk) | 0/407 | 0/407 | 0/407 | 0/407 | 0/407 | 0/407 | 0/407
Other Adverse Events (participants affected / at risk) | 0/407 | 0/407 | 0/407 | 0/407 | 0/407 | 0/407 | 0/407

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-22): https://cdn.clinicaltrials.gov/large-docs/69/NCT05393869/Prot_SAP_000.pdf